CLINICAL TRIAL: NCT03553940
Title: A Phase I Trial to Evaluate the Safety and Immunogenicity of an Influenza Vaccination Strategy Including a H3N2 M2SR Prime Followed by a Seasonal Quadrivalent Inactivated Vaccine Boost in a Pediatric Population 9-17 Years Old
Brief Title: H3N2 M2SR in Pediatric Population
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-0012; HHSN272201300021I
Record Dates: First submitted 2018-05-31; First posted 2018-06-12 (Actual); Results first posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-03-01

CONDITIONS: Influenza; Influenza Immunisation
Keywords: H3N2 M2SR Prime; Immunogenicity; Influenza; Pediatric Population; QIV; Safety; Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): A single dose of monovalent live attenuated influenza H3N2 M2SR vaccine (M2SR) administered intranasally on Day 1, and a single dose of licensed quadrivalent influenza vaccine (QIV) administered intramuscularly on Day 92. N=25
  Interventions: Biological: Influenza Virus Monovalent A/H3N2/Bris 10 M2SR Live Vaccine; Biological: Quadrivalent MDCK Inactivated Influenza Vaccine
- Arm 2 (Placebo Comparator): A single dose of Placebo administered intranasally on Day 1, and a single dose of licensed QIV administered intramuscularly on Day 92. N=25
  Interventions: Other: Placebo; Biological: Quadrivalent MDCK Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: Influenza Virus Monovalent A/H3N2/Bris 10 M2SR Live Vaccine — Live monovalent influenza A/H3N2-based M2SR (M2 defective Single Replication vaccine), comprised of 5 out of 8 gene segments on the donor virus influenza A/Puerto Rica/8/34. HA and NA derive from an A/Brisbane/10/2007-like virus. Administered intranasally as s single dose.
  Arms: Arm 1
Other: Placebo — H3N2 M2SR vaccine placebo (normal saline). Administered intranasally as a single dose.
  Arms: Arm 2
Biological: Quadrivalent MDCK Inactivated Influenza Vaccine — A quadrivalent cell culture inactivated vaccine (ccIV4) is an inactivated subunit influenza vaccine prepared from virus propagated in Madin Darby Canine Kidney (MDCK) cells indicated for the prevention of influenza disease caused by influenza virus subtypes A and type B contained in the vaccine. Administered intramuscularly as a single dose.

SUMMARY:
This is a Phase I double-blind, randomized, placebo-controlled study in 50 healthy adolescents and children, 9-17 years of age, inclusive, who are in good health and meet all eligibility criteria. This clinical trial is designed to assess the safety and immunogenicity of a prime-boost regimen of H3N2 M2SR intranasal influenza vaccine (manufactured by FluGen) followed by licensed inactivated Quadrivalent Influenza Vaccine (QIV) boost administered intramuscularly Subjects will be enrolled in one of two groups in a 1:1 ratio. Arm 1 will receive one dose of M2SR intranasally on Day 1 and one dose of QIV on Day 92. Arm 2 will receive one dose of placebo (saline) intranasally on Day 1, and one dose of QIV on Day 92. Study duration will be approximately 28 months with patient participation duration approximately 13 months. The primary study objective is to assess the safety and reactogenicity of a monovalent live attenuated influenza H3N2 M2SR vaccine.

DETAILED DESCRIPTION:
This is a Phase I double-blind, randomized, placebo-controlled study in 50 healthy adolescents and children, 9-17 years of age, inclusive, who are in good health and meet all eligibility criteria. This clinical trial is designed to assess the safety and immunogenicity of a prime-boost regimen of H3N2 M2SR intranasal influenza vaccine (manufactured by FluGen) followed by licensed inactivated Quadrivalent Influenza Vaccine (QIV) boost administered intramuscularly. Subjects will be enrolled in one of two groups in a 1:1 ratio. Arm 1 will receive one dose of M2SR intranasally on Day 1 and one dose of QIV on Day 92. Arm 2 will receive one dose of placebo (saline) intranasally on Day 1, and one dose of QIV on Day 92. Study duration will be approximately 28 months with patient participation duration approximately 13 months. The primary study objective is to assess the safety and reactogenicity of a monovalent live attenuated influenza H3N2 M2SR vaccine. The secondary study objectives are to identify circulating and mucosal antibody responses induced by H3N2 M2SR vaccination and to identify cellular immune responses induced by H3N2 M2SR vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Parent(s)/legal guardian(s) must provide written informed consent prior to initiation of any study procedures, and subject must provide assent.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Are males or non-pregnant females, 9-17 years old, inclusive at the time of enrollment.
4. Are in good health*.

   *As determined by medical history and physical examination to evaluate acute or currently ongoing chronic medical diagnoses or conditions, defined as those that have been present for at least 90 days, which would affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions should be stable for the last 60 days (no hospitalizations, ER, or urgent care for condition and no adverse symptoms that need medical intervention). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis or condition in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided there was no deterioration in the subject's chronic medical condition that necessitated a medication change, and there is no additional risk to the subject or interference with the evaluation of responses to study vaccination. Note: Low dose topical steroids, herbals, vitamins, and supplements are permitted.
5. Oral temperature is less than 100.0 degrees Fahrenheit.
6. For female adolescent of child-bearing potential* must agree to correctly use an acceptable method of contraception** from 30 days prior to vaccination until 30 days after the last study vaccination.

   *Defined by the onset of menses, and not sterilized via tubal ligation, bilateral oophorectomy, hysterectomy, or successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating.

   **Includes non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with a vasectomized partner, and correct use of male condoms with the use of applied spermicide, intrauterine devices, NuvaRing(R), and licensed hormonal methods such as implants, injectables, contraceptive patches or oral contraceptives ("the pill"). Method of contraception will be captured on the appropriate data collection form.
7. Female adolescent of childbearing potential must have a negative urine pregnancy test within 24 hours prior to study vaccination.
8. Males who are sexually active with a female of childbearing potential must agree not to father a child for 30 days after receipt of the first study vaccination.
9. Agrees not to participate in another clinical trial during the study period.
10. Agrees not to donate blood or blood products to a blood bank for 12 months after receiving the investigational vaccine.
11. Weight = / > 34 kg or 75 pounds.
12. Hemoglobin = / > 11.5 g/dL.
13. Hematocrit > 35%.
14. Ferritin level = / > 15 ng/mL.
15. Parent/legal guardian must provide consent to future use of stored samples.

Exclusion Criteria:

1. Have an acute illness*, as determined by the site PI or appropriate sub-investigator, within 72 hours prior to each study vaccination.

   *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
2. Have any medical disease or condition that, in the opinion of the site PI or appropriate sub-investigator, is a contraindication to study participation*.

   *Including acute or chronic medical disease or condition, defined as persisting for at least 90 days, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this study.
3. Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
4. Have known active neoplastic disease or a history of any hematologic malignancy. Non-melanoma skin cancers that are not active are permitted.
5. Have known HIV, hepatitis B, or hepatitis C infection.
6. Have a history of severe reactions following previous immunization with licensed or unlicensed influenza vaccines.
7. History of anatomic disorder of the nares or nasopharynx (Deviated septum is allowed).
8. History of chronic sinus infections.
9. Have a history of Guillain-Barre Syndrome.
10. Have a history of alcohol or drug abuse prior to study vaccination.
11. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
12. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others prior to study vaccination.
13. Have taken oral and/or nasal corticosteroids of any dose within 30 days prior to each study vaccination or plan to take in the 30 days following the first study vaccination.
14. Have taken high-dose*,** inhaled corticosteroids within 30 days (prior to study vaccination).

    *High-dose defined as per age as using inhaled high dose per reference chart.

    **https://www.nhlbi.nih.gov/files/docs/guidelines/asthma_org.pdf.
15. Use of aspirin or salicylate-containing products 30 days prior to the first vaccination.
16. Recurring or active wheezing or diagnosis of asthma, or history of significant wheezing*.

    *Medically significant wheezing: defined as wheezing on physical exam plus sign of respiratory distress (tachypnea, retractions, or dyspnea), hypoxemia (O2 saturation < 95%), or new bronchodilator prescription, or use of daily bronchodilator therapy (not on an "as needed" basis).
17. Received any licensed live or inactivated vaccine within 30 days prior to or plan to receive any licensed live or inactivated vaccine within 30 days after each study vaccination.
18. Received any influenza vaccine (inactivated or live) within 6 months prior to the first study vaccination and until the end of the study.
19. Received immunoglobulin or other blood products within 6 months prior to study vaccination.
20. Received an experimental agent* within 30 days prior to the first study vaccination, or expects to receive an experimental agent** during the 12-month trial-reporting period.

    *Including vaccine, drug, biologic, device, blood product, or medication.

    **Other than from participation in this study.
21. Are participating or plan to participate in another clinical trial with an interventional agent* that will be received during the 12-month trial-reporting period.

    *Including agent (licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication) during the 12-month study period.
22. Prior history of H3N2 actual or potential exposure or infection prior to the first study vaccination, or receipt of experimental vaccines within the past year prior to the first study vaccine.
23. Female adolescent subject who is breastfeeding or plans to breastfeed at any given time from the first study vaccination until 30 days after the last study vaccination.
24. Blood donation within 30 days prior to the study vaccination through 30 days after the last blood drawn for this study.
25. Have signs or symptoms that could confound or confuse assessment of study vaccine reactogenicity*.

    *The study vaccination should be postponed/deferred until signs or symptoms have resolved and if within the acceptable protocol-specified window for that visit.
26. Have received any antiviral drug within 3 days of study vaccination.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis University - Center for Vaccine Development, St Louis, Missouri, United States

REFERENCES:
- [Derived] Taaffe J, Ostrowsky JT, Mott J, Goldin S, Friede M, Gsell P, Chadwick C. Advancing influenza vaccines: A review of next-generation candidates and their potential for global health impact. Vaccine. 2024 Dec 2;42(26):126408. doi: 10.1016/j.vaccine.2024.126408. Epub 2024 Oct 5. PMID 39369576

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy males and non-pregnant females between 9 and 17 years old, inclusively. They were recruited from the community at large around the clinic site. Participants were enrolled between 15AUG2018 and 20SEP2019.
Groups:
- M2SR: A single dose of monovalent live attenuated influenza H3N2 M2SR vaccine (M2SR) administered intranasally on Day 1, and a single dose of licensed quadrivalent influenza vaccine (QIV) administered intramuscularly on Day 92.
  Influenza Virus Monovalent A/H3N2/Bris 10 M2SR Live Vaccine: Live monovalent influenza A/H3N2-based M2SR (M2 defective Single Replication vaccine), comprised of 5 out of 8 gene segments on the donor virus influenza A/Puerto Rico/8/34. HA and NA derive from an A/Brisbane/10/2007-like virus. Administered intranasally as a single dose.
  Quadrivalent MDCK Inactivated Influenza Vaccine: A quadrivalent cell culture inactivated vaccine (ccIV4) is an inactivated subunit influenza vaccine prepared from virus propagated in Madin Darby Canine Kidney (MDCK) cells indicated for the prevention of influenza disease caused by influenza virus subtypes A and B contained in the vaccine. Administered intramuscularly as a single dose.
- Placebo: A single dose of Placebo administered intranasally on Day 1, and a single dose of licensed QIV administered intramuscularly on Day 92.
  Placebo: H3N2 M2SR vaccine placebo (normal saline). Administered intranasally as a single dose.
  Quadrivalent MDCK Inactivated Influenza Vaccine: A quadrivalent cell culture inactivated vaccine (ccIV4) is an inactivated subunit influenza vaccine prepared from virus propagated in Madin Darby Canine Kidney (MDCK) cells indicated for the prevention of influenza disease caused by influenza virus subtypes A and B contained in the vaccine. Administered intramuscularly as a single dose.
Period: Overall Study
Arm/Group | M2SR | Placebo
Started | 22 | 21
Completed | 22 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all enrolled participants.
Groups:
- M2SR: A single dose of monovalent live attenuated influenza H3N2 M2SR vaccine (M2SR) administered intranasally on Day 1, and a single dose of licensed quadrivalent influenza vaccine (QIV) administered intramuscularly on Day 92.
- Placebo: A single dose of Placebo administered intranasally on Day 1, and a single dose of licensed QIV administered intramuscularly on Day 92.
- Total: Total of all reporting groups
Arm/Group | M2SR | Placebo | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (1.8) | 12.9 (2.2) | 13.3 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 21 | 18 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 19 | 39
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: Adverse Events of Special Interest (AESIs) included medically significant wheezing and otitis media. AESIs were collected from receipt of the first study vaccination through 3 months after first vaccination.
Time Frame: Day 1 through Day 92
Population: The Safety population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
Participants | 0 | 0

2. Primary Outcome: Number of Participants With New Onset Chronic Medical Conditions (NOCMCs)
Description: Participants were queried at each visit for the occurrence of new onset chronic medical conditions (NOCMCs). NOCMCs were collected from receipt of the first study vaccination through 3 months after first vaccination.
Time Frame: Day 1 through Day 92
Population: The Safety population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect.
Time Frame: Day 1 through Day 366
Population: The Safety population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Solicited Reactogenicity
Description: Reactogenicity assessments included an assessment of solicited AEs occurring from the time of first study vaccination through 7 days after first vaccination. For upper respiratory symptoms, this included an assessment of runny nose, stuffy nose/ congestion, sneezing, nasal pain/irritation/nasal dryness, nasal bleeding/epistaxis, sinus pressure/pain, sore throat/sore/scratchy, itchy or painful throat, cough, and trouble breathing/shortness of breath. For general systemic symptoms, this included an assessment of reactions including fever, feverishness (chills/shivering/sweating), fatigue (tiredness), malaise, myalgia (body aches/muscular pain), arthralgia (joint pain), headache, flushing, decreased activity, decreased appetite, abdominal pain, nausea, vomiting, diarrhea, eye pruritus, eye redness (conjunctivitis), allergy, and wheezing.
Time Frame: Day 1 through Day 8
Population: The Safety population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
Participants
  Upper Respiratory Symptoms | 5 | 7
  Systemic Symptoms | 11 | 10

5. Primary Outcome: Number of Participants With Unsolicited Non-Serious Adverse Events
Description: Adverse events were defined as any untoward medical occurrence in a participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Non-serious AEs were collected from the time of first study vaccination through 21 days after first vaccination. Adverse events were MedDRA coded and are summarized by MedDRA System Organ Class (SOC).
Time Frame: Day 1 through Day 22
Population: The Safety population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
Participants | 6 | 5

6. Secondary Outcome: Frequency of Conserved Internal Viral Protein-specific Spot Forming Cells
Description: Blood was collected for ELISpot assays conducted with a peptide library consisting of conserved immunogenic peptides of internal flu virus proteins as the antigen . Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). Peripheral blood mononuclear cells (PBMCs) were harvested and retained from each whole blood collection. The geometric mean of each sample's replicate results was calculated from available results using spot forming cells per 3x10^5 peripheral blood mononuclear cells (SFC/3x10^5 PBMCs).
Time Frame: Day 1 through Day 113
Population: The Modified Intent-to-Treat (mITT) population includes all participants who received at least one dose of study vaccine and contributed both pre- and at least one post-study vaccination venous blood samples for which valid results were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: SFC/3x10^5 PBMCs
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
SFC/3x10^5 PBMCs
  Day 1 | 17.2 [12.6 to 23.3] | 23.0 [12.8 to 41.2]
  Day 8 | 24.1 [17.3 to 33.5] | 23.5 [13.7 to 40.2]
  Day 22 | 24.5 [17.1 to 35.0] | 20.2 [11.2 to 36.2]
  Day 57 | 16.2 [11.3 to 23.4] | 21.4 [13.5 to 33.8]
  Day 92: number analyzed (Participants) | 15 | 17
  Day 92 | 16.3 [9.7 to 27.3] | 17.0 [9.6 to 30.1]
  Day 113: number analyzed (Participants) | 15 | 17
  Day 113 | 20.8 [13.4 to 32.2] | 22.3 [12.6 to 39.6]

7. Secondary Outcome: Frequency of Influenza H3 HA-specific Spot Forming Cells for the H3N2 M2SR-like Virus A/Brisbane/10/2007
Description: Blood was collected for ELISpot assays conducted with H3N2 M2SR-like virus A/Brisbane/10/2007 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). Peripheral blood mononuclear cells (PBMCs) were harvested and retained from each whole blood collection. The geometric mean of each sample's replicate results was calculated from available results using spot forming cells per 3x10^5 peripheral blood mononuclear cells (SFC/3x10^5 PBMCs).
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: SFC/3x10^5 PBMCs
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
SFC/3x10^5 PBMCs
  Day 1 | 37.5 [22.1 to 63.6] | 50.2 [33.7 to 74.6]
  Day 8 | 48.9 [26.0 to 91.8] | 59.0 [35.5 to 98.1]
  Day 22 | 65.8 [35.3 to 122.6] | 46.3 [21.6 to 99.2]
  Day 57 | 41.8 [22.8 to 76.9] | 45.1 [26.5 to 76.8]
  Day 92: number analyzed (Participants) | 15 | 17
  Day 92 | 30.2 [14.2 to 64.2] | 32.2 [15.6 to 66.3]
  Day 113: number analyzed (Participants) | 15 | 17
  Day 113 | 34.0 [18.4 to 62.7] | 50.4 [29.3 to 86.5]

8. Secondary Outcome: Frequency of Influenza H3 HA-specific Spot Forming Cells for the H3N2 QIV-like Virus A/North Carolina/04/2016
Description: Blood was collected for ELISpot assays conducted with H3N2 QIV-like virus A/North Carolina/04/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). Peripheral blood mononuclear cells (PBMCs) were harvested and retained from each whole blood collection. The geometric mean of each sample's replicate results was calculated from available results using spot forming cells per 3x10^5 peripheral blood mononuclear cells (SFC/3x10^5 PBMCs).
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: SFC/3x10^5 PBMCs
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
SFC/3x10^5 PBMCs
  Day 1 | 30.7 [17.7 to 53.4] | 42.5 [27.0 to 66.9]
  Day 8 | 39.7 [22.1 to 71.6] | 45.1 [27.5 to 74.0]
  Day 22 | 49.5 [26.0 to 94.2] | 40.0 [19.0 to 84.0]
  Day 57 | 30.0 [15.7 to 57.2] | 40.5 [24.7 to 66.5]
  Day 92: number analyzed (Participants) | 14 | 17
  Day 92 | 18.5 [7.5 to 45.4] | 30.0 [15.0 to 60.1]
  Day 113: number analyzed (Participants) | 15 | 17
  Day 113 | 25.2 [13.2 to 47.9] | 39.8 [23.6 to 67.0]

9. Secondary Outcome: Frequency of Influenza H3 HA-specific Spot Forming Cells for the H3N2 QIV-like Virus A/Singapore/INFIMH-16-0019/2016
Description: Blood was collected for ELISpot assays conducted with H3N2 QIV-like virus A/Singapore/INFIMH-16-0019/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). Peripheral blood mononuclear cells (PBMCs) were harvested and retained from each whole blood collection. The geometric mean of each sample's replicate results was calculated from available results using spot forming cells per 3x10^5 peripheral blood mononuclear cells (SFC/3x10^5 PBMCs).
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: SFC/3x10^5 PBMCs
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
SFC/3x10^5 PBMCs
  Day 1 | 31.5 [18.9 to 52.5] | 42.1 [27.8 to 63.6]
  Day 8 | 40.5 [23.9 to 68.8] | 46.0 [28.4 to 74.5]
  Day 22 | 50.9 [26.5 to 97.8] | 40.2 [19.4 to 83.3]
  Day 57 | 35.3 [21.0 to 59.6] | 39.2 [24.1 to 63.9]
  Day 92: number analyzed (Participants) | 14 | 17
  Day 92 | 26.2 [13.8 to 49.6] | 29.6 [16.0 to 54.9]
  Day 113: number analyzed (Participants) | 15 | 17
  Day 113 | 25.2 [14.0 to 45.1] | 40.7 [23.7 to 69.9]

10. Secondary Outcome: Frequency of Influenza H3 HA-specific Spot Forming Cells for the H3N2 QIV-like Virus A/Kansas/14/2017
Description: Blood was collected for ELISpot assays conducted with H3N2 QIV-like virus A/Kansas/14/2017 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). Peripheral blood mononuclear cells (PBMCs) were harvested and retained from each whole blood collection. The geometric mean of each sample's replicate results was calculated from available results using spot forming cells per 3x10^5 peripheral blood mononuclear cells (SFC/3x10^5 PBMCs).
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: SFC/3x10^5 PBMCs
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
SFC/3x10^5 PBMCs
  Day 1 | 5.3 [3.8 to 7.4] | 5.3 [3.5 to 7.9]
  Day 8 | 7.1 [4.9 to 10.3] | 6.0 [3.6 to 10.0]
  Day 22 | 5.4 [3.6 to 8.1] | 6.6 [3.9 to 11.3]
  Day 57 | 4.7 [3.4 to 6.3] | 5.2 [3.4 to 7.9]
  Day 92: number analyzed (Participants) | 14 | 17
  Day 92 | 4.3 [2.9 to 6.5] | 4.3 [2.7 to 6.8]
  Day 113: number analyzed (Participants) | 15 | 17
  Day 113 | 4.9 [3.2 to 7.4] | 6.4 [3.9 to 10.7]

11. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Nasal Secretory Immunoglobulin A (sIgA) Responses Directed Against the H3N2 M2SR-like Virus A/Brisbane/10/2007
Description: Nasal swabs were collected for secretory immunoglobulin A (sIgA) assays conducted with H3N2 M2SR-like virus A/Brisbane/10/2007 as the antigen. Collection took place Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Geometric mean fold rise (GMFR) was calculated by dividing each post-baseline geometric mean titer by baseline geometric mean titer. The GMFR across samples was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
ratio
  Day 8 | 1.1 [0.4 to 2.9] | 1.2 [0.5 to 3.3]
  Day 22 | 1.3 [0.4 to 4.2] | 1.9 [1.0 to 3.4]
  Day 57 | 0.8 [0.2 to 3.1] | 1.9 [0.7 to 5.1]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 1.3 [0.5 to 3.7] | 1.4 [0.7 to 3.1]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 1.8 [0.6 to 5.6] | 4.9 [2.3 to 10.6]

12. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Nasal Secretory Immunoglobulin A (sIgA) Responses Directed Against the H3N2 M2SR-like Virus A/Brisbane/10/2007 Normalized to Total sIgA
Description: Nasal swabs were collected for secretory immunoglobulin A (sIgA) assays conducted with H3N2 M2SR-like virus A/Brisbane/10/2007 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Results were normalized to total sIgA by dividing each geometric mean titer by total sIgA concentration (ng/mL). Geometric mean fold rise (GMFR) was calculated by dividing each post-baseline normalized geometric mean titer by baseline normalized geometric mean titer. The GMFR across samples was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
ratio
  Day 8 | 1.9 [0.9 to 4.1] | 1.6 [0.8 to 3.5]
  Day 22 | 1.9 [0.9 to 4.1] | 1.3 [0.8 to 1.9]
  Day 57 | 1.0 [0.4 to 2.4] | 1.2 [0.5 to 2.5]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 1.3 [0.6 to 2.6] | 0.8 [0.3 to 2.0]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 1.1 [0.7 to 1.8] | 1.6 [0.7 to 3.7]

13. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Nasal Secretory Immunoglobulin A (sIgA) Responses Directed Against the H3N2 QIV-like Virus A/North Carolina/04/2016
Description: Nasal swabs were collected for secretory immunoglobulin A (sIgA) assays conducted with H3N2 QIV-like virus A/North Carolina/04/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Geometric mean fold rise (GMFR) was calculated by dividing each post-baseline geometric mean titer by baseline geometric mean titer. The GMFR across samples was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
ratio
  Day 8 | 0.7 [0.2 to 1.9] | 0.7 [0.3 to 1.9]
  Day 22 | 0.8 [0.2 to 2.6] | 1.2 [0.7 to 2.0]
  Day 57 | 0.7 [0.2 to 2.0] | 1.1 [0.4 to 3.1]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 1.0 [0.5 to 2.4] | 1.1 [0.4 to 2.7]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 1.6 [0.5 to 5.2] | 2.5 [0.9 to 6.9]

14. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Nasal Secretory Immunoglobulin A (sIgA) Responses Directed Against the H3N2 QIV-like Virus A/North Carolina/04/2016 Normalized to Total sIgA
Description: Nasal swabs were collected for secretory immunoglobulin A (sIgA) assays conducted with H3N2 QIV-like virus A/North Carolina/04/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Results were normalized to total sIgA by dividing each geometric mean titer by total sIgA concentration (ng/mL). Geometric mean fold rise (GMFR) was calculated by dividing each post-baseline normalized geometric mean titer by baseline normalized geometric mean titer. The GMFR across samples was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
ratio
  Day 8 | 1.2 [0.6 to 2.6] | 1.0 [0.5 to 1.9]
  Day 22 | 1.1 [0.6 to 2.0] | 0.8 [0.5 to 1.5]
  Day 57 | 0.8 [0.4 to 1.7] | 0.7 [0.4 to 1.3]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 1.0 [0.7 to 1.6] | 0.6 [0.4 to 1.1]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 1.0 [0.6 to 1.7] | 0.8 [0.4 to 1.5]

15. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Nasal Secretory Immunoglobulin A (sIgA) Responses Directed Against the H3N2 QIV-like Virus A/Singapore/INFIMH-16-0019/2016
Description: Nasal swabs were collected for secretory immunoglobulin A (sIgA) assays conducted with H3N2 QIV-like virus A/Singapore/INFIMH-16-0019/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Geometric mean fold rise (GMFR) was calculated by dividing each post-baseline geometric mean titer by baseline geometric mean titer. The GMFR across samples was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
ratio
  Day 8 | 0.7 [0.3 to 1.5] | 0.5 [0.2 to 1.0]
  Day 22 | 1.3 [0.6 to 3.1] | 1.1 [0.6 to 2.3]
  Day 57 | 0.6 [0.3 to 1.1] | 0.8 [0.4 to 1.6]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 0.8 [0.4 to 1.8] | 0.5 [0.2 to 1.2]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 0.9 [0.3 to 2.7] | 0.9 [0.4 to 2.2]

16. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Nasal Secretory Immunoglobulin A (sIgA) Responses Directed Against the H3N2 QIV-like Virus A/Singapore/INFIMH-16-0019/2016 Normalized to Total sIgA
Description: Nasal swabs were collected for secretory immunoglobulin A (sIgA) assays conducted with H3N2 QIV-like virus A/Singapore/INFIMH-16-0019/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Results were normalized to total sIgA by dividing each geometric mean titer by total sIgA concentration (ng/mL). Geometric mean fold rise (GMFR) was calculated by dividing each post-baseline normalized geometric mean titer by baseline normalized geometric mean titer. The GMFR across samples was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
ratio
  Day 8 | 1.2 [0.6 to 2.5] | 0.7 [0.3 to 1.6]
  Day 22 | 1.9 [0.8 to 4.4] | 0.8 [0.4 to 1.5]
  Day 57 | 0.7 [0.3 to 1.8] | 0.5 [0.2 to 1.2]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 0.8 [0.4 to 1.7] | 0.3 [0.1 to 0.8]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 0.6 [0.2 to 1.7] | 0.3 [0.1 to 0.8]

17. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Nasal Secretory Immunoglobulin A (sIgA) Responses Directed Against the H3N2 QIV-like Virus A/Kansas/14/2017
Description: Nasal swabs were collected for secretory immunoglobulin A (sIgA) assays conducted with H3N2 QIV-like virus A/Kansas/14/2017 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Geometric mean fold rise (GMFR) was calculated by dividing each post-baseline geometric mean titer by baseline geometric mean titer. The GMFR across samples was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
ratio
  Day 8 | 0.6 [0.2 to 1.7] | 0.5 [0.2 to 1.3]
  Day 22 | 1.1 [0.4 to 2.8] | 1.3 [0.5 to 3.4]
  Day 57 | 0.6 [0.2 to 1.7] | 1.2 [0.4 to 3.6]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 1.4 [0.6 to 3.5] | 1.1 [0.5 to 2.3]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 1.3 [0.3 to 5.4] | 3.8 [1.4 to 10.2]

18. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Nasal Secretory Immunoglobulin A (sIgA) Responses Directed Against the H3N2 QIV-like Virus A/Kansas/14/2017 Normalized to Total sIgA
Description: Nasal swabs were collected for secretory immunoglobulin A (sIgA) assays conducted with H3N2 QIV-like virus A/Kansas/14/2017 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Results were normalized to total sIgA by dividing each geometric mean titer by total sIgA concentration (ng/mL). Geometric mean fold rise (GMFR) was calculated by dividing each post-baseline normalized geometric mean titer by baseline normalized geometric mean titer. The GMFR across samples was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
ratio
  Day 8 | 1.1 [0.6 to 2.1] | 0.7 [0.3 to 1.5]
  Day 22 | 1.6 [0.8 to 3.3] | 0.8 [0.4 to 1.9]
  Day 57 | 0.7 [0.3 to 1.7] | 0.8 [0.4 to 1.7]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 1.4 [0.8 to 2.3] | 0.6 [0.3 to 1.3]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 0.9 [0.4 to 2.0] | 1.2 [0.6 to 2.6]

19. Secondary Outcome: Geometric Mean Titer (GMT) of Nasal Secretory Immunoglobulin A (sIgA) Responses Directed Against the H3N2 M2SR-like Virus A/Brisbane/10/2007
Description: Nasal swabs were collected for secretory immunoglobulin A (sIgA) assays conducted with H3N2 M2SR-like virus A/Brisbane/10/2007 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
titer
  Day 1 | 17.3 [7.0 to 42.4] | 8.4 [3.9 to 18.1]
  Day 8 | 18.9 [7.4 to 48.3] | 10.3 [3.8 to 28.2]
  Day 22 | 22.9 [8.5 to 61.5] | 15.9 [8.9 to 28.5]
  Day 57 | 13.8 [5.4 to 35.3] | 16.0 [6.1 to 42.0]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 21.2 [10.2 to 44.0] | 12.0 [5.7 to 25.4]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 28.4 [11.5 to 70.1] | 41.2 [15.6 to 109.2]

20. Secondary Outcome: Geometric Mean Titer (GMT) of Nasal Secretory Immunoglobulin A (sIgA) Responses Directed Against the H3N2 M2SR-like Virus A/Brisbane/10/2007 Normalized to Total sIgA
Description: Nasal swabs were collected for secretory immunoglobulin A (sIgA) assays conducted with H3N2 M2SR-like virus A/Brisbane/10/2007 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Results were normalized to total sIgA by dividing each geometric mean titer by total sIgA concentration (ng/ml). The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer per ng/mL sIgA
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
titer per ng/mL sIgA
  Day 1 | 1.5 [0.6 to 3.4] | 1.4 [0.7 to 3.0]
  Day 8 | 2.9 [1.7 to 4.9] | 2.3 [1.2 to 4.7]
  Day 22 | 2.8 [1.5 to 5.4] | 1.8 [0.9 to 3.6]
  Day 57 | 1.5 [0.6 to 3.5] | 1.7 [0.7 to 3.7]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 1.8 [0.9 to 3.9] | 1.2 [0.4 to 3.3]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 1.6 [0.8 to 3.2] | 2.3 [0.9 to 5.8]

21. Secondary Outcome: Geometric Mean Titer (GMT) of Nasal Secretory Immunoglobulin A (sIgA) Responses Directed Against the H3N2 QIV-like Virus A/North Carolina/04/2016
Description: Nasal swabs were collected for secretory immunoglobulin A (sIgA) assays conducted with H3N2 QIV-like virus A/North Carolina/04/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
titer
  Day 1 | 25.5 [10.9 to 59.4] | 16.7 [6.2 to 45.0]
  Day 8 | 17.5 [7.6 to 40.1] | 12.5 [4.9 to 31.7]
  Day 22 | 19.5 [7.3 to 52.5] | 20.4 [9.8 to 42.3]
  Day 57 | 16.9 [7.3 to 39.0] | 18.6 [6.9 to 49.9]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 25.8 [13.2 to 50.6] | 18.2 [8.1 to 41.2]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 38.1 [16.6 to 87.2] | 41.3 [15.4 to 110.8]

22. Secondary Outcome: Geometric Mean Titer (GMT) of Nasal Secretory Immunoglobulin A (sIgA) Responses Directed Against the H3N2 QIV-like Virus A/North Carolina/04/2016 Normalized to Total sIgA
Description: Nasal swabs were collected for secretory immunoglobulin A (sIgA) assays conducted with H3N2 QIV-like virus A/North Carolina/04/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Results were normalized to total sIgA by dividing each geometric mean titer by total sIgA concentration (ng/ml). The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer per ng/mL sIgA
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
titer per ng/mL sIgA
  Day 1 | 2.2 [1.2 to 4.0] | 2.8 [1.1 to 7.0]
  Day 8 | 2.7 [1.5 to 4.8] | 2.8 [1.4 to 5.7]
  Day 22 | 2.4 [1.4 to 4.3] | 2.3 [1.0 to 5.4]
  Day 57 | 1.8 [0.9 to 3.7] | 1.9 [0.8 to 4.5]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 2.2 [1.3 to 3.9] | 1.8 [0.8 to 4.4]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 2.1 [1.2 to 3.6] | 2.3 [0.9 to 5.9]

23. Secondary Outcome: Geometric Mean Titer (GMT) of Nasal Secretory Immunoglobulin A (sIgA) Responses Directed Against the H3N2 QIV-like Virus A/Singapore/INFIMH-16-0019/2016
Description: Nasal swabs were collected for secretory immunoglobulin A (sIgA) assays conducted with H3N2 QIV-like virus A/Singapore/INFIMH-16-0019/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
titer
  Day 1 | 29.7 [15.0 to 58.6] | 26.1 [10.9 to 62.1]
  Day 8 | 20.2 [9.3 to 44.0] | 12.8 [5.4 to 30.4]
  Day 22 | 39.0 [18.0 to 84.4] | 29.8 [14.2 to 62.4]
  Day 57 | 16.7 [8.6 to 32.7] | 21.4 [9.6 to 47.5]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 24.6 [12.3 to 49.1] | 14.3 [6.8 to 30.0]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 25.7 [11.9 to 55.6] | 23.0 [8.9 to 59.2]

24. Secondary Outcome: Geometric Mean Titer (GMT) of Nasal Secretory Immunoglobulin A (sIgA) Responses Directed Against the H3N2 QIV-like Virus A/Singapore/INFIMH-16-0019/2016 Normalized to Total sIgA
Description: Nasal swabs were collected for secretory immunoglobulin A (sIgA) assays conducted with H3N2 QIV-like virus A/Singapore/INFIMH-16-0019/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Results were normalized to total sIgA by dividing each geometric mean titer by total sIgA concentration (ng/ml). The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer per ng/mL sIgA
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
titer per ng/mL sIgA
  Day 1 | 2.6 [1.3 to 5.1] | 4.4 [1.7 to 11.6]
  Day 8 | 3.1 [1.4 to 6.9] | 2.9 [1.1 to 7.5]
  Day 22 | 4.8 [2.7 to 8.8] | 3.4 [1.3 to 8.9]
  Day 57 | 1.8 [0.7 to 4.5] | 2.2 [0.8 to 6.1]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 2.1 [1.0 to 4.5] | 1.4 [0.6 to 3.6]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 1.4 [0.5 to 3.6] | 1.3 [0.4 to 4.4]

25. Secondary Outcome: Geometric Mean Titer (GMT) of Nasal Secretory Immunoglobulin A (sIgA) Responses Directed Against the H3N2 QIV-like Virus A/Kansas/14/2017
Description: Nasal swabs were collected for secretory immunoglobulin A (sIgA) assays conducted with H3N2 QIV-like virus A/Kansas/14/2017 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
titer
  Day 1 | 17.1 [6.8 to 43.1] | 9.9 [3.9 to 25.5]
  Day 8 | 10.8 [4.2 to 27.6] | 5.0 [2.0 to 12.6]
  Day 22 | 19.0 [8.3 to 43.5] | 12.5 [4.4 to 35.7]
  Day 57 | 9.4 [4.1 to 21.5] | 12.4 [5.4 to 28.5]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 23.2 [12.2 to 44.3] | 10.7 [5.9 to 19.4]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 23.0 [9.5 to 55.7] | 38.0 [18.4 to 78.5]

26. Secondary Outcome: Geometric Mean Titer (GMT) of Nasal Secretory Immunoglobulin A (sIgA) Responses Directed Against the H3N2 QIV-like Virus A/Kansas/14/2017 Normalized to Total sIgA
Description: Nasal swabs were collected for secretory immunoglobulin A (sIgA) assays conducted with H3N2 QIV-like virus A/Kansas/14/2017 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Results were normalized to total sIgA by dividing each geometric mean titer by total sIgA concentration (ng/ml). The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer per ng/mL sIgA
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
titer per ng/mL sIgA
  Day 1 | 1.5 [0.8 to 2.7] | 1.7 [0.7 to 4.1]
  Day 8 | 1.6 [0.8 to 3.3] | 1.1 [0.5 to 2.4]
  Day 22 | 2.4 [1.2 to 4.6] | 1.4 [0.6 to 3.6]
  Day 57 | 1.0 [0.4 to 2.4] | 1.3 [0.7 to 2.5]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 2.0 [1.1 to 3.5] | 1.1 [0.5 to 2.1]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 1.3 [0.6 to 2.7] | 2.1 [1.0 to 4.3]

27. Secondary Outcome: Hemagglutination Inhibition (HAI) Antibody Geometric Mean Fold Rise (GMFR) to the H3N2 M2SR-like Virus A/Brisbane/10/2007
Description: Blood was collected for HAI assays conducted with H3N2 M2SR-like virus A/Brisbane/10/2007 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Geometric mean fold rise (GMFR) was calculated by dividing each post-baseline geometric mean titer by baseline geometric mean titer. The GMFR across samples was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
ratio
  Day 8 | 1.0 [1.0 to 1.1] | 1.0 [0.9 to 1.0]
  Day 22 | 1.2 [1.0 to 1.3] | 1.0 [0.9 to 1.0]
  Day 57 | 1.1 [0.9 to 1.3] | 1.0 [0.9 to 1.1]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 1.1 [1.0 to 1.3] | 1.0 [0.9 to 1.0]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 1.9 [1.3 to 2.9] | 1.9 [1.3 to 2.9]

28. Secondary Outcome: Hemagglutination Inhibition (HAI) Antibody Geometric Mean Fold Rise (GMFR) to the H3N2 QIV-like Virus A/North Carolina/04/2016
Description: Blood was collected for HAI assays conducted with H3N2 QIV-like virus A/North Carolina/04/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Geometric mean fold rise (GMFR) was calculated by dividing each post-baseline geometric mean titer by baseline geometric mean titer. The GMFR across samples was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
ratio
  Day 8 | 1.0 [0.9 to 1.0] | 1.0 [NA to NA] — Not calculable due to insufficient variability.
  Day 22 | 1.0 [0.9 to 1.0] | 1.0 [NA to NA] — Not calculable due to insufficient variability.
  Day 57 | 1.0 [0.9 to 1.0] | 1.0 [NA to NA] — Not calculable due to insufficient variability.
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 1.0 [NA to NA] — Not calculable due to insufficient variability. | 1.0 [NA to NA] — Not calculable due to insufficient variability.
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 2.3 [1.8 to 2.8] | 3.2 [2.4 to 4.2]

29. Secondary Outcome: Hemagglutination Inhibition (HAI) Antibody Geometric Mean Fold Rise (GMFR) to the H3N2 QIV-like Virus A/Singapore/INFIMH-16-0019/2016
Description: Blood was collected for HAI assays conducted with H3N2 QIV-like virus A/Singapore/INFIMH-16-0019/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Geometric mean fold rise (GMFR) was calculated by dividing each post-baseline geometric mean titer by baseline geometric mean titer. The GMFR across samples was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
ratio
  Day 8 | 1.0 [NA to NA] — Not calculable due to insufficient variability. | 0.9 [0.9 to 1.0]
  Day 22 | 1.0 [1.0 to 1.1] | 0.9 [0.9 to 1.0]
  Day 57 | 1.0 [1.0 to 1.1] | 0.9 [0.9 to 1.0]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 1.0 [0.9 to 1.1] | 0.9 [0.8 to 1.0]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 2.3 [1.4 to 3.8] | 2.4 [1.7 to 3.6]

30. Secondary Outcome: Hemagglutination Inhibition (HAI) Antibody Geometric Mean Fold Rise (GMFR) to the H3N2 QIV-like Virus A/Kansas/14/2017
Description: Blood was collected for HAI assays conducted with H3N2 QIV-like virus A/Kansas/14/2017 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Geometric mean fold rise (GMFR) was calculated by dividing each post-baseline geometric mean titer by baseline geometric mean titer. The GMFR across samples was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
ratio
  Day 8 | 1.0 [NA to NA] — Not calculable due to insufficient variability. | 1.0 [0.9 to 1.1]
  Day 22 | 1.0 [NA to NA] — Not calculable due to insufficient variability. | 0.9 [0.9 to 1.0]
  Day 57 | 1.0 [1.0 to 1.1] | 1.0 [0.9 to 1.2]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 1.0 [1.0 to 1.1] | 1.0 [0.9 to 1.1]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 3.2 [1.7 to 5.8] | 4.4 [2.5 to 7.9]

31. Secondary Outcome: Hemagglutination Inhibition (HAI) Antibody Geometric Mean Titers (GMTs) to the H3N2 M2SR-like Virus A/Brisbane/10/2007
Description: Blood was collected for HAI assays conducted with H3N2 M2SR-like virus A/Brisbane/10/2007 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
titer
  Day 1 | 93.6 [55.7 to 157.3] | 67.8 [42.5 to 108.2]
  Day 8 | 96.6 [57.4 to 162.7] | 65.6 [41.9 to 102.7]
  Day 22 | 109.6 [68.4 to 175.7] | 65.6 [41.9 to 102.7]
  Day 57 | 102.9 [66.3 to 159.9] | 67.8 [43.0 to 107.0]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 107.7 [68.5 to 169.3] | 65.6 [41.9 to 102.7]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 188.7 [133.7 to 266.3] | 131.3 [87.9 to 196.0]

32. Secondary Outcome: Hemagglutination Inhibition (HAI) Antibody Geometric Mean Titers (GMTs) to the H3N2 QIV-like Virus A/North Carolina/04/2016
Description: Blood was collected for HAI assays conducted with H3N2 QIV-like virus A/North Carolina/04/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
titer
  Day 1 | 14.1 [11.1 to 18.1] | 13.5 [10.2 to 17.7]
  Day 8 | 13.7 [10.5 to 17.8] | 13.5 [10.2 to 17.7]
  Day 22 | 13.7 [10.5 to 17.8] | 13.5 [10.2 to 17.7]
  Day 57 | 13.7 [10.5 to 17.8] | 13.5 [10.2 to 17.7]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 14.4 [11.1 to 18.6] | 13.5 [10.2 to 17.7]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 31.7 [24.2 to 41.6] | 42.7 [28.7 to 63.6]

33. Secondary Outcome: Hemagglutination Inhibition (HAI) Antibody Geometric Mean Titers (GMTs) to the H3N2 QIV-like Virus A/Singapore/INFIMH-16-0019/2016
Description: Blood was collected for HAI assays conducted with H3N2 QIV-like virus A/Singapore/INFIMH-16-0019/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
titer
  Day 1 | 96.6 [61.8 to 151.1] | 88.3 [61.4 to 127.1]
  Day 8 | 96.6 [61.8 to 151.1] | 82.7 [58.1 to 117.6]
  Day 22 | 99.7 [64.3 to 154.7] | 82.7 [58.1 to 117.6]
  Day 57 | 99.7 [64.3 to 154.7] | 82.7 [58.1 to 117.6]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 94.4 [60.5 to 147.3] | 80.0 [55.8 to 114.6]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 230.0 [153.2 to 345.5] | 215.3 [151.2 to 306.7]

34. Secondary Outcome: Hemagglutination Inhibition (HAI) Antibody Geometric Mean Titers (GMTs) to the H3N2 QIV-like Virus A/Kansas/14/2017
Description: Blood was collected for HAI assays conducted with H3N2 QIV-like virus A/Kansas/14/2017 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
titer
  Day 1 | 25.7 [18.2 to 36.5] | 25.2 [17.5 to 36.3]
  Day 8 | 25.7 [18.2 to 36.5] | 25.2 [17.3 to 36.8]
  Day 22 | 25.7 [18.2 to 36.5] | 23.6 [17.0 to 32.8]
  Day 57 | 26.6 [19.0 to 37.2] | 25.2 [17.3 to 36.8]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 26.0 [18.3 to 37.0] | 25.2 [17.7 to 35.8]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 85.5 [44.1 to 165.5] | 111.3 [62.9 to 196.8]

35. Secondary Outcome: Neutralizing Antibody Geometric Mean Fold Rise (GMFR) to the H3N2 M2SR-like Virus A/Brisbane/10/2007
Description: Blood was collected for Neutralizing assays conducted with H3N2 M2SR-like virus A/Brisbane/10/2007 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Geometric mean fold rise (GMFR) was calculated by dividing each post-baseline geometric mean titer by baseline geometric mean titer. The GMFR across samples was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
ratio
  Day 8 | 1.0 [0.9 to 1.2] | 1.0 [0.9 to 1.1]
  Day 22 | 1.1 [0.9 to 1.4] | 1.0 [0.9 to 1.1]
  Day 57 | 1.2 [1.0 to 1.4] | 0.9 [0.8 to 1.0]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 1.1 [0.9 to 1.3] | 0.9 [0.8 to 1.1]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 1.8 [1.2 to 2.6] | 1.9 [1.3 to 2.8]

36. Secondary Outcome: Neutralizing Antibody Geometric Mean Fold Rise (GMFR) to the H3N2 QIV-like Virus A/North Carolina/04/2016
Description: Blood was collected for Neutralizing assays conducted with H3N2 QIV-like virus A/North Carolina/04/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Geometric mean fold rise (GMFR) was calculated by dividing each post-baseline geometric mean titer by baseline geometric mean titer. The GMFR across samples was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
ratio
  Day 8 | 1.1 [0.9 to 1.2] | 1.0 [0.9 to 1.1]
  Day 22 | 1.0 [0.9 to 1.2] | 1.0 [0.9 to 1.1]
  Day 57 | 1.0 [0.9 to 1.2] | 1.0 [0.9 to 1.1]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 1.0 [0.9 to 1.2] | 0.9 [0.8 to 1.0]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 2.6 [1.9 to 3.8] | 4.5 [2.9 to 6.8]

37. Secondary Outcome: Neutralizing Antibody Geometric Mean Fold Rise (GMFR) to the H3N2 QIV-like Virus A/Singapore/INFIMH-16-0019/2016
Description: Blood was collected for Neutralizing assays conducted with H3N2 QIV-like virus A/Singapore/INFIMH-16-0019/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Geometric mean fold rise (GMFR) was calculated by dividing each post-baseline geometric mean titer by baseline geometric mean titer. The GMFR across samples was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
ratio
  Day 8 | 1.0 [0.9 to 1.2] | 1.0 [0.9 to 1.1]
  Day 22 | 1.0 [0.9 to 1.1] | 1.0 [0.9 to 1.0]
  Day 57 | 1.0 [0.9 to 1.2] | 0.9 [0.9 to 1.0]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 1.0 [0.9 to 1.1] | 1.0 [0.9 to 1.1]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 2.9 [1.6 to 5.3] | 2.9 [2.0 to 4.3]

38. Secondary Outcome: Neutralizing Antibody Geometric Mean Fold Rise (GMFR) to the H3N2 QIV-like Virus A/Kansas/14/2017
Description: Blood was collected for Neutralizing assays conducted with H3N2 QIV-like virus A/Kansas/14/2017 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Geometric mean fold rise (GMFR) was calculated by dividing each post-baseline geometric mean titer by baseline geometric mean titer. The GMFR across samples was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
ratio
  Day 8 | 1.0 [0.8 to 1.1] | 1.1 [0.9 to 1.3]
  Day 22 | 1.0 [0.8 to 1.1] | 1.1 [0.9 to 1.3]
  Day 57 | 0.9 [0.8 to 1.0] | 0.9 [0.8 to 1.0]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 0.9 [0.7 to 1.1] | 1.0 [0.9 to 1.1]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 3.0 [1.6 to 5.4] | 4.7 [2.6 to 8.5]

39. Secondary Outcome: Neutralizing Antibody Geometric Mean Titers (GMTs) to the H3N2 M2SR-like Virus A/Brisbane/10/2007
Description: Blood was collected for Neutralizing assays conducted with H3N2 M2SR-like virus A/Brisbane/10/2007 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
titer
  Day 1 | 1374.0 [818.4 to 2307.0] | 1178.6 [754.0 to 1842.2]
  Day 8 | 1418.0 [847.3 to 2373.1] | 1159.3 [707.2 to 1900.4]
  Day 22 | 1558.6 [1036.3 to 2344.1] | 1188.4 [755.6 to 1869.0]
  Day 57 | 1595.9 [1035.2 to 2460.1] | 1076.3 [679.5 to 1704.9]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 1509.7 [978.3 to 2329.6] | 1112.5 [703.5 to 1759.3]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 2497.4 [1658.5 to 3760.6] | 2206.7 [1405.3 to 3465.1]

40. Secondary Outcome: Neutralizing Antibody Geometric Mean Titers (GMTs) to the H3N2 QIV-like Virus A/North Carolina/04/2016
Description: Blood was collected for Neutralizing assays conducted with H3N2 QIV-like virus A/North Carolina/04/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
titer
  Day 1 | 70.5 [47.2 to 105.5] | 83.4 [52.0 to 133.7]
  Day 8 | 74.5 [48.9 to 113.5] | 80.0 [47.9 to 133.5]
  Day 22 | 72.8 [47.1 to 112.5] | 84.1 [51.0 to 138.6]
  Day 57 | 71.1 [44.8 to 112.7] | 81.3 [50.9 to 129.9]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 75.5 [50.0 to 114.1] | 77.4 [47.2 to 126.8]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 185.6 [108.6 to 317.2] | 371.2 [221.7 to 621.7]

41. Secondary Outcome: Neutralizing Antibody Geometric Mean Titers (GMTs) to the H3N2 QIV-like Virus A/Singapore/INFIMH-16-0019/2016
Description: Blood was collected for Neutralizing assays conducted with H3N2 QIV-like virus A/Singapore/INFIMH-16-0019/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
titer
  Day 1 | 726.0 [428.1 to 1231.1] | 700.8 [511.4 to 960.4]
  Day 8 | 755.1 [438.3 to 1301.0] | 706.6 [508.2 to 982.5]
  Day 22 | 726.0 [442.9 to 1189.8] | 667.0 [476.9 to 932.8]
  Day 57 | 755.1 [489.1 to 1165.8] | 661.5 [470.5 to 930.0]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 700.8 [413.7 to 1187.2] | 683.7 [488.6 to 956.7]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 2206.7 [1390.0 to 3503.0] | 2031.9 [1530.0 to 2698.3]

42. Secondary Outcome: Neutralizing Antibody Geometric Mean Titers (GMTs) to the H3N2 QIV-like Virus A/Kansas/14/2017
Description: Blood was collected for Neutralizing assays conducted with H3N2 QIV-like virus A/Kansas/14/2017 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The geometric mean titer (GMT) across samples was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
titer
  Day 1 | 196.4 [126.6 to 304.6] | 165.4 [113.5 to 240.9]
  Day 8 | 190.3 [122.3 to 295.9] | 176.7 [115.6 to 269.9]
  Day 22 | 190.3 [135.7 to 266.7] | 182.6 [122.3 to 272.5]
  Day 57 | 175.9 [114.7 to 269.6] | 152.3 [97.7 to 237.4]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 182.6 [126.3 to 263.9] | 162.7 [109.3 to 242.0]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 619.2 [331.5 to 1156.7] | 780.2 [411.4 to 1479.6]

43. Secondary Outcome: Percentage of Participants Achieving a Serum Hemagglutination Inhibition (HAI) Antibody Titer of >= 1:40 Against the H3N2 M2SR-like Virus A/Brisbane/10/2007
Description: Blood was collected for HAI assays conducted with H3N2 M2SR-like virus A/Brisbane/10/2007 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The percentage of participants with HAI geometric mean titer >= 1:40 was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
percentage of participants
  Day 1 | 82 [61 to 94] | 86 [65 to 96]
  Day 8 | 82 [61 to 94] | 86 [65 to 96]
  Day 22 | 86 [67 to 96] | 86 [65 to 96]
  Day 57 | 86 [67 to 96] | 86 [65 to 96]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 86 [65 to 96] | 86 [65 to 96]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 100 [85 to 100] | 95 [77 to 100]

44. Secondary Outcome: Percentage of Participants Achieving a Serum Hemagglutination Inhibition (HAI) Antibody Titer of >= 1:40 Against the H3N2 QIV-like Virus A/North Carolina/04/2016
Description: Blood was collected for HAI assays conducted with H3N2 QIV-like virus A/North Carolina/04/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The percentage of participants with HAI geometric mean titer >= 1:40 was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
percentage of participants
  Day 1 | 9 [2 to 29] | 5 [0 to 23]
  Day 8 | 9 [2 to 29] | 5 [0 to 23]
  Day 22 | 9 [2 to 29] | 5 [0 to 23]
  Day 57 | 9 [2 to 29] | 5 [0 to 23]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 10 [2 to 30] | 5 [0 to 23]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 57 [35 to 77] | 67 [45 to 85]

45. Secondary Outcome: Percentage of Participants Achieving a Serum Hemagglutination Inhibition (HAI) Antibody Titer of >= 1:40 Against the H3N2 QIV-like Virus A/Singapore/INFIMH-16-0019/2016
Description: Blood was collected for HAI assays conducted with H3N2 QIV-like virus A/Singapore/INFIMH-16-0019/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The percentage of participants with HAI geometric mean titer >= 1:40 was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
percentage of participants
  Day 1 | 91 [71 to 98] | 95 [77 to 100]
  Day 8 | 91 [71 to 98] | 95 [77 to 100]
  Day 22 | 91 [71 to 98] | 95 [77 to 100]
  Day 57 | 91 [71 to 98] | 95 [77 to 100]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 90 [70 to 98] | 95 [77 to 100]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 95 [77 to 100] | 100 [85 to 100]

46. Secondary Outcome: Percentage of Participants Achieving a Serum Hemagglutination Inhibition (HAI) Antibody Titer of >= 1:40 Against the H3N2 QIV-like Virus A/Kansas/14/2017
Description: Blood was collected for HAI assays conducted with H3N2 QIV-like virus A/Kansas/14/2017 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The percentage of participants with HAI geometric mean titer >= 1:40 was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
percentage of participants
  Day 1 | 41 [22 to 62] | 38 [20 to 60]
  Day 8 | 41 [22 to 62] | 33 [15 to 55]
  Day 22 | 41 [22 to 62] | 33 [15 to 55]
  Day 57 | 41 [22 to 62] | 33 [15 to 55]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 38 [20 to 60] | 33 [15 to 55]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 86 [65 to 96] | 90 [70 to 98]

47. Secondary Outcome: Percentage of Participants Achieving a Serum Neutralizing Antibody Titer of >= 1:40 Against the H3N2 M2SR-like Virus A/Brisbane/10/2007
Description: Blood was collected for Neutralizing assays conducted with H3N2 M2SR-like virus A/Brisbane/10/2007 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The percentage of participants with HAI geometric mean titer >= 1:40 was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
percentage of participants
  Day 1 | 100 [85 to 100] | 100 [85 to 100]
  Day 8 | 100 [85 to 100] | 100 [85 to 100]
  Day 22 | 100 [85 to 100] | 100 [85 to 100]
  Day 57 | 100 [85 to 100] | 100 [85 to 100]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 100 [85 to 100] | 100 [85 to 100]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 100 [85 to 100] | 100 [85 to 100]

48. Secondary Outcome: Percentage of Participants Achieving a Serum Neutralizing Antibody Titer of >= 1:40 Against the H3N2 QIV-like Virus A/North Carolina/04/2016
Description: Blood was collected for Neutralizing assays conducted with H3N2 QIV-like virus A/North Carolina/04/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The percentage of participants with HAI geometric mean titer >= 1:40 was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
percentage of participants
  Day 1 | 77 [55 to 91] | 81 [60 to 93]
  Day 8 | 82 [61 to 94] | 81 [60 to 93]
  Day 22 | 77 [55 to 91] | 81 [60 to 93]
  Day 57 | 77 [55 to 91] | 81 [60 to 93]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 81 [60 to 93] | 81 [60 to 93]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 100 [85 to 100] | 100 [85 to 100]

49. Secondary Outcome: Percentage of Participants Achieving a Serum Neutralizing Antibody Titer of >= 1:40 Against the H3N2 QIV-like Virus A/Singapore/INFIMH-16-0019/2016
Description: Blood was collected for Neutralizing assays conducted with H3N2 QIV-like virus A/Singapore/INFIMH-16-0019/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The percentage of participants with HAI geometric mean titer >= 1:40 was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
percentage of participants
  Day 1 | 95 [78 to 100] | 100 [85 to 100]
  Day 8 | 95 [78 to 100] | 100 [85 to 100]
  Day 22 | 95 [78 to 100] | 100 [85 to 100]
  Day 57 | 100 [85 to 100] | 100 [85 to 100]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 95 [77 to 100] | 100 [85 to 100]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 100 [85 to 100] | 100 [85 to 100]

50. Secondary Outcome: Percentage of Participants Achieving a Serum Neutralizing Antibody Titer of >= 1:40 Against the H3N2 QIV-like Virus A/Kansas/14/2017
Description: Blood was collected for Neutralizing assays conducted with H3N2 QIV-like virus A/Kansas/14/2017 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. The percentage of participants with HAI geometric mean titer >= 1:40 was calculated within each study arm and analysis time point.
Time Frame: Day 1 through Day 113
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
percentage of participants
  Day 1 | 95 [78 to 100] | 100 [85 to 100]
  Day 8 | 95 [78 to 100] | 100 [85 to 100]
  Day 22 | 100 [85 to 100] | 100 [85 to 100]
  Day 57 | 95 [78 to 100] | 95 [77 to 100]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 95 [77 to 100] | 95 [77 to 100]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 100 [85 to 100] | 100 [85 to 100]

51. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Seroconversion Against the H3N2 M2SR-like Virus A/Brisbane/10/2007
Description: Blood was collected for HAI assays conducted with H3N2 M2SR-like virus A/Brisbane/10/2007 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Seroconversion is defined as either a pre-vaccination geometric mean titer (GMT) < 1:10 and a post-vaccination GMT >= 1:40, or a pre-vaccination GMT >= 1:10 and a minimum 4-fold rise in post-vaccination GMT. The percentage of participants achieving seroconversion was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
percentage of participants
  Day 8 | 0 [0 to 15] | 0 [0 to 15]
  Day 22 | 0 [0 to 15] | 0 [0 to 15]
  Day 57 | 0 [0 to 15] | 0 [0 to 15]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 0 [0 to 15] | 0 [0 to 15]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 24 [10 to 46] | 19 [7 to 40]

52. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Seroconversion Against the H3N2 QIV-like Virus A/North Carolina/04/2016
Description: Blood was collected for HAI assays conducted with H3N2 QIV-like virus A/North Carolina/04/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Seroconversion is defined as either a pre-vaccination geometric mean titer (GMT) < 1:10 and a post-vaccination GMT >= 1:40, or a pre-vaccination GMT >= 1:10 and a minimum 4-fold rise in post-vaccination GMT. The percentage of participants achieving seroconversion was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
percentage of participants
  Day 8 | 0 [0 to 15] | 0 [0 to 15]
  Day 22 | 0 [0 to 15] | 0 [0 to 15]
  Day 57 | 0 [0 to 15] | 0 [0 to 15]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 0 [0 to 15] | 0 [0 to 15]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 24 [10 to 46] | 62 [40 to 80]

53. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Seroconversion Against the H3N2 QIV-like Virus A/Singapore/INFIMH-16-0019/2016
Description: Blood was collected for HAI assays conducted with H3N2 QIV-like virus A/Singapore/INFIMH-16-0019/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Seroconversion is defined as either a pre-vaccination geometric mean titer (GMT) < 1:10 and a post-vaccination GMT >= 1:40, or a pre-vaccination GMT >= 1:10 and a minimum 4-fold rise in post-vaccination GMT. The percentage of participants achieving seroconversion was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
percentage of participants
  Day 8 | 0 [0 to 15] | 0 [0 to 15]
  Day 22 | 0 [0 to 15] | 0 [0 to 15]
  Day 57 | 0 [0 to 15] | 0 [0 to 15]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 0 [0 to 15] | 0 [0 to 15]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 24 [10 to 46] | 33 [15 to 55]

54. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Seroconversion Against the H3N2 QIV-like Virus A/Kansas/14/2017
Description: Blood was collected for HAI assays conducted with H3N2 QIV-like virus A/Kansas/14/2017 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Seroconversion is defined as either a pre-vaccination geometric mean titer (GMT) < 1:10 and a post-vaccination GMT >= 1:40, or a pre-vaccination GMT >= 1:10 and a minimum 4-fold rise in post-vaccination GMT. The percentage of participants achieving seroconversion was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
percentage of participants
  Day 8 | 0 [0 to 15] | 0 [0 to 15]
  Day 22 | 0 [0 to 15] | 0 [0 to 15]
  Day 57 | 0 [0 to 15] | 0 [0 to 15]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 0 [0 to 15] | 0 [0 to 15]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 43 [23 to 65] | 52 [30 to 72]

55. Secondary Outcome: Percentage of Participants Achieving Neutralizing Antibody Seroconversion Against the H3N2 M2SR-like Virus A/Brisbane/10/2007
Description: Blood was collected for Neutralizing assays conducted with H3N2 M2SR-like virus A/Brisbane/10/2007 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Seroconversion is defined as either a pre-vaccination geometric mean titer (GMT) < 1:10 and a post-vaccination GMT >= 1:40, or a pre-vaccination GMT >= 1:10 and a minimum 4-fold rise in post-vaccination GMT. The percentage of participants achieving seroconversion was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
percentage of participants
  Day 8 | 0 [0 to 15] | 0 [0 to 15]
  Day 22 | 0 [0 to 15] | 0 [0 to 15]
  Day 57 | 0 [0 to 15] | 0 [0 to 15]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 0 [0 to 15] | 0 [0 to 15]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 24 [10 to 46] | 19 [7 to 40]

56. Secondary Outcome: Percentage of Participants Achieving Neutralizing Antibody Seroconversion Against the H3N2 QIV-like Virus A/North Carolina/04/2016
Description: Blood was collected for Neutralizing assays conducted with H3N2 QIV-like virus A/North Carolina/04/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Seroconversion is defined as either a pre-vaccination geometric mean titer (GMT) < 1:10 and a post-vaccination GMT >= 1:40, or a pre-vaccination GMT >= 1:10 and a minimum 4-fold rise in post-vaccination GMT. The percentage of participants achieving seroconversion was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
percentage of participants
  Day 8 | 0 [0 to 15] | 0 [0 to 15]
  Day 22 | 0 [0 to 15] | 0 [0 to 15]
  Day 57 | 0 [0 to 15] | 0 [0 to 15]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 0 [0 to 15] | 0 [0 to 15]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 33 [15 to 55] | 62 [40 to 80]

57. Secondary Outcome: Percentage of Participants Achieving Neutralizing Antibody Seroconversion Against the H3N2 QIV-like Virus A/Singapore/INFIMH-16-0019/2016
Description: Blood was collected for Neutralizing assays conducted with H3N2 QIV-like virus A/Singapore/INFIMH-16-0019/2016 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Seroconversion is defined as either a pre-vaccination geometric mean titer (GMT) < 1:10 and a post-vaccination GMT >= 1:40, or a pre-vaccination GMT >= 1:10 and a minimum 4-fold rise in post-vaccination GMT. The percentage of participants achieving seroconversion was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
percentage of participants
  Day 8 | 0 [0 to 15] | 0 [0 to 15]
  Day 22 | 0 [0 to 15] | 0 [0 to 15]
  Day 57 | 0 [0 to 15] | 0 [0 to 15]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 0 [0 to 15] | 0 [0 to 15]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 38 [20 to 60] | 43 [23 to 65]

58. Secondary Outcome: Percentage of Participants Achieving Neutralizing Antibody Seroconversion Against the H3N2 QIV-like Virus A/Kansas/14/2017
Description: Blood was collected for Neutralizing assays conducted with H3N2 QIV-like virus A/Kansas/14/2017 as the antigen. Collection took place on Day 1 (pre-vaccination), Days 8, 22, and 57 after first vaccination, immediately prior to second vaccination (Day 92), and 21 days after second vaccination (Day 113). The geometric mean of each sample's replicate results was calculated from available results. Seroconversion is defined as either a pre-vaccination geometric mean titer (GMT) < 1:10 and a post-vaccination GMT >= 1:40, or a pre-vaccination GMT >= 1:10 and a minimum 4-fold rise in post-vaccination GMT. The percentage of participants achieving seroconversion was calculated within each study arm and analysis time point.
Time Frame: Day 8 through Day 113
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M2SR | Placebo
Number analyzed (Participants) | 22 | 21
percentage of participants
  Day 8 | 0 [0 to 15] | 0 [0 to 15]
  Day 22 | 0 [0 to 15] | 0 [0 to 15]
  Day 57 | 0 [0 to 15] | 0 [0 to 15]
  Day 92: number analyzed (Participants) | 21 | 21
  Day 92 | 0 [0 to 15] | 0 [0 to 15]
  Day 113: number analyzed (Participants) | 21 | 21
  Day 113 | 43 [23 to 65] | 48 [28 to 70]

ADVERSE EVENTS:
Time Frame: Solicited reactogenicity events were reported from the time of experimental (first) study vaccination through Day 8 after vaccination. Unsolicited non-serious AEs were reported from the time of the first study vaccination through Day 22 after the first study vaccination. SAEs were reported from the time of the first study vaccination through Day 366 after the first vaccination. AESIs and NOCMCs were reported from the time of first study vaccination through Day 92 after first study vaccination.
Arm/Group | M2SR | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 11/22 | 17/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M2SR (N=22) | Placebo (N=21)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 5 (5) | 4 (4)
Malaise (General disorders) | 3 (3) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 3 (3)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 8 (8) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Flushing (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT03553940/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/40/NCT03553940/SAP_001.pdf